CLINICAL TRIAL: NCT01467466
Title: CSP #578 - Prevention of Serious Adverse Events Following Angiography (PRESERVE)
Brief Title: Prevention of Serious Adverse Events Following Angiography
Acronym: PRESERVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: The George Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 578; 1011387 (Other Grant/Funding Number: National Health and Medical Research Council)
Record Dates: First submitted 2011-10-26; First posted 2011-11-08 (Estimated); Results first posted 2018-11-09 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Acute Renal Failure; Kidney Disease; Coronary Artery Disease
Keywords: renal; cardiovascular; kidney; heart; clinical trial; double-blind; multi-site trial; randomized; drug treatment; IV solutions; antioxidant
MeSH Terms: conditions — Acute Kidney Injury; Kidney Diseases; Coronary Artery Disease | interventions — Sodium Chloride; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Saline & oral placebo (Active Comparator): IV isotonic saline and oral placebo drug capsule
  Interventions: Drug: IV isotonic saline; Drug: Placebo
- Saline & oral N-acetylcysteine (Active Comparator): IV isotonic saline and oral N-acetylcysteine drug capsule
  Interventions: Drug: IV isotonic saline; Drug: N-acetylcysteine
- Bicarbonate & oral placebo (Active Comparator): IV isotonic bicarbonate and oral placebo drug capsule
  Interventions: Drug: IV isotonic bicarbonate; Drug: Placebo
- Bicarbonate & oral N-acetylcysteine (Active Comparator): IV isotonic bicarbonate and oral N-acetylcysteine drug capsule
  Interventions: Drug: IV isotonic bicarbonate; Drug: N-acetylcysteine

INTERVENTIONS:
Drug: IV isotonic saline — The investigators will administer 3 ml/kg of isotonic saline over 1 hour at an infusion rate of not less than 1 mL/kg per hour and not more than 3 mL/kg per hour prior to the angiographic procedure, 1-1.5ml/kg per hour during angiography, and 6 ml/kg of isotonic saline over 4 hours following the procedure at an infusion rate of not less than 1 mL/kg per hour and not more than 1.5 mL/kg per hour. Providers will retain discretion to administer larger volumes of isotonic saline (up to a maximum of 12 mL/kg) over durations of up to 12 hours pre and 12 hours post-procedure.
  Arms: Saline & oral N-acetylcysteine; Saline & oral placebo
Drug: IV isotonic bicarbonate — The investigators will administer 3 ml/kg of isotonic bicarbonate over 1 hour at an infusion rate of not less than 1 mL/kg per hour and not more than 3 mL/kg per hour prior to the angiographic procedure, 1-1.5ml/kg per hour during angiography, and 6 ml/kg of isotonic bicarbonate over 4 hours following the procedure at an infusion rate of not less than 1 mL/kg per hour and not more than 1.5 mL/kg per hour. Providers will retain discretion to administer larger volumes of isotonic bicarbonate (up to a maximum of 12 mL/kg) over durations of up to 12 hours pre and 12 hours post-procedure.
  Arms: Bicarbonate & oral N-acetylcysteine; Bicarbonate & oral placebo
Drug: N-acetylcysteine — NAC will be administered at a dose of 1200mg orally 1 hour prior to angiography, 1 hour following the procedure, and then twice daily for the next 4 days.
  Other Names: NAC
  Arms: Bicarbonate & oral N-acetylcysteine; Saline & oral N-acetylcysteine
Drug: Placebo — A placebo study drug capsule will be administered orally 1 hour prior to angiography, 1 hour following the procedure, and then twice daily for the next 4 days.
  Arms: Bicarbonate & oral placebo; Saline & oral placebo

SUMMARY:
The purpose of this research study is to compare the effectiveness of intravenous isotonic sodium bicarbonate with intravenous isotonic sodium chloride and oral N-acetylcysteine (NAC) with oral placebo for the prevention of serious adverse outcomes following angiographic procedures in high-risk patients.

DETAILED DESCRIPTION:
The intravascular administration of iodinated contrast media for diagnostic imaging is a common cause of acute kidney injury (AKI) and a leading cause of iatrogenic renal disease. Contrast-induced AKI is associated with serious adverse outcomes including death, need for dialysis, prolonged hospitalization, and acceleration in the rate of progression of underlying chronic kidney disease. The benefit of IV isotonic bicarbonate compared to IV isotonic saline and of N-acetylcysteine for the prevention of contrast-induced AKI and associated adverse outcomes remains unclear. The purpose of this trial is to compare the effectiveness of IV isotonic sodium bicarbonate with IV isotonic sodium chloride and oral NAC with placebo for the prevention of serious adverse outcomes in 7,680 high-risk patients scheduled to undergo coronary or non-coronary angiography. Using a 2 x 2 factorial design, patients will be randomized to receive: 1) either peri-procedural IV isotonic sodium bicarbonate or peri-procedural IV isotonic saline and 2) either oral NAC or oral placebo prior to and for 5 days following the angiographic procedure. The primary study endpoint is a composite outcome comprised of death, need for acute dialysis, or persistent decline in kidney function within 90 days following the index angiogram.

ELIGIBILITY:
Inclusion Criteria:

* Planned elective or urgent coronary or non-coronary angiography with iodinated contrast media in which it is anticipated that there will be an interval of 3 hours between the identification of the indication for angiography and the time of the planned procedure.
* Pre-angiography eGFR <60 ml/min/1.73 m2 with diabetes mellitus or pre-angiography eGFR <45 ml/min/1.73 m2 with or without diabetes mellitus
* Ability to provide informed consent

Exclusion Criteria:

* Stage 5 chronic kidney disease (CKD) (eGFR <15 mL/min/1.73 m2)
* Currently receiving hemodialysis, peritoneal dialysis, continuous renal replacement therapy, or sustained low efficiency dialysis (SLED)
* Unstable baseline serum creatinine (SCr) (if known) at the time of angiography defined by an increase in SCr of 25% over the 3 days prior to angiography
* Decompensated heart failure requiring any of the following therapies at the time of angiography:

  * IV milrinone, amrinone, dobutamine, or nesiritide
  * Isolated ultrafiltration therapy
  * Intra-aortic balloon pump
* Emergent angiography procedures defined as an anticipated duration of <3 hours between the identification of the indication for angiography and the time of the planned procedure.
* Receipt of intravascular iodinated contrast within the 5 days preceding angiography
* Receipt of oral or IV NAC within the 48 hours preceding angiography
* Known allergy to N-acetylcysteine (NAC)
* Known anaphylactic allergy to iodinated contrast media
* Prisoner
* Age <18 years
* Pregnancy
* Ongoing participation in an unapproved concurrent interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5177 (Actual)
Dates: Start 2013-10-07 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven D. Weisbord, MD MSc, Study Chair — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (54):
- United States (35):
  - Southern Arizona VA Health Care System, Tucson, Tucson, Arizona
  - Central Arkansas VHS John L. McClellan Memorial Veterans Hospital, Little Rock, AR, Little Rock, Arkansas
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Bay Pines VA Healthcare System, Pay Pines, FL, Bay Pines, Florida
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Charlie Norwood VA Medical Center, Augusta, GA, Augusta, Georgia
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - VA Boston Healthcare System West Roxbury Campus, West Roxbury, MA, West Roxbury, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Kansas City VA Medical Center, Kansas City, MO, Kansas City, Missouri
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Dayton VA Medical Center, Dayton, OH, Dayton, Ohio
  - Oklahoma City VA Medical Center, Oklahoma City, OK, Oklahoma City, Oklahoma
  - Portland VA Medical Center, Portland, OR, Portland, Oregon
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - Memphis VA Medical Center, Memphis, TN, Memphis, Tennessee
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia
  - Salem VA Medical Center, Salem, VA, Salem, Virginia
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington
- Australia (13):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Concord Hospital, Concord, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - St. George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Northern Health, Epping, Victoria
  - Austin Health, Heidelberg, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Malaysia (3):
  - University of Malaya Medical Center, Kuala Lumpur, Kuala Lumpur
  - Penang Hospital, George Town, Pulau Pinang
  - Hospital Serdang, Sepang, Selangor
- New Zealand (3):
  - Auckland City Hospital, Auckland, Auckland
  - Taranaki Base Hospital, Westown, New Plymouth
  - Wellington Hospital, Newtown, Wellington Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weisbord SD, Gallagher M, Jneid H, Garcia S, Cass A, Thwin SS, Conner TA, Chertow GM, Bhatt DL, Shunk K, Parikh CR, McFalls EO, Brophy M, Ferguson R, Wu H, Androsenko M, Myles J, Kaufman J, Palevsky PM; PRESERVE Trial Group. Outcomes after Angiography with Sodium Bicarbonate and Acetylcysteine. N Engl J Med. 2018 Feb 15;378(7):603-614. doi: 10.1056/NEJMoa1710933. Epub 2017 Nov 12. PMID 29130810

RESULTS

PARTICIPANT FLOW:
Groups:
- Saline & oral N-acetylcysteine: IV isotonic saline and oral N-acetylcysteine (NAC) drug capsule
  IV isotonic saline: The investigators will administer 3 ml/kg of isotonic saline over 1 hour at an infusion rate of not less than 1 mL/kg per hour and not more than 3 mL/kg per hour prior to the angiographic procedure, 1-1.5ml/kg per hour during angiography, and 6 ml/kg of isotonic saline over 4 hours following the procedure at an infusion rate of not less than 1 mL/kg per hour and not more than 1.5 mL/kg per hour. Providers will retain discretion to administer larger volumes of isotonic saline (up to a maximum of 12 mL/kg) over durations of up to 12 hours pre and 12 hours post-procedure.
  N-acetylcysteine: NAC will be administered at a dose of 1200mg orally 1 hour prior to angiography, 1 hour following the procedure, and then twice daily for the next 4 days.
Period: Overall Study
Arm/Group | Saline & oral placebo | Saline & oral N-acetylcysteine | Bicarbonate & oral placebo | Bicarbonate & oral N-acetylcysteine
Started | 1300 | 1292 | 1294 | 1291
Completed | 1191 | 1188 | 1190 | 1203
Not Completed | 109 | 104 | 104 | 88
Not completed — Withdrawal by Subject | 15 | 18 | 13 | 11
Not completed — Revoked Consent Prior To Procedure | 10 | 9 | 15 | 5
Not completed — Procedure Cancelled | 46 | 45 | 25 | 29
Not completed — No Endpoint Blood Draw | 38 | 32 | 51 | 43

BASELINE CHARACTERISTICS:
Population: A total of 5,177 participants were randomized into this trial. 4,993 participants completed baseline activities and summary information is provided below. A total of 4,772 participants were assessed for the primary outcome, which accounts for the discrepancy in numbers reported between baseline and outcome sections in this submission.
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline & oral placebo | Saline & oral N-acetylcysteine | Bicarbonate & oral placebo | Bicarbonate & oral N-acetylcysteine | Total
Number analyzed (Participants) | 1244 | 1238 | 1254 | 1257 | 4993
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.6 (8.4) | 69.8 (8.3) | 69.6 (8.3) | 70.2 (8.0) | 69.8 (8.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 86 | 75 | 87 | 73 | 321
  Sex: Male | 1157 | 1163 | 1167 | 1184 | 4671
  Sex: Unknown/Not Stated | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 11 | 7 | 9 | 8 | 35
  Race: Asian | 64 | 58 | 69 | 65 | 256
  Race: Native Hawaiian or Other Pacific Islander | 19 | 10 | 16 | 17 | 62
  Race: Black or AFrican American | 141 | 158 | 150 | 121 | 570
  Race: White | 971 | 967 | 962 | 993 | 3893
  Race: Indigenous Austrailian | 1 | 1 | 0 | 2 | 4
  Race: More than one race | 31 | 37 | 43 | 50 | 161
  Race: Unknown or Not Reported | 6 | 0 | 5 | 1 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Spanish, Hispanic or Latino | 1190 | 1198 | 1179 | 1197 | 4764
  Ethnicity: Mexican, Mexican American, or Chicano | 17 | 9 | 27 | 20 | 73
  Ethnicity: Puerto Rican | 5 | 3 | 1 | 3 | 12
  Ethnicity: Cuban | 0 | 1 | 0 | 0 | 1
  Ethnicity: Other Spanish Hispanic, or Latino | 21 | 16 | 31 | 27 | 95
  Ethnicity: Chose Not to Answer | 11 | 11 | 16 | 10 | 48
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 45 | 45 | 44 | 45 | 179
  United States | 1068 | 1054 | 1068 | 1077 | 4267
  Malaysia | 56 | 57 | 59 | 58 | 230
  Australia | 75 | 82 | 83 | 77 | 317

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious, Adverse, Patient-Centered Events, Including Death, Need for Acute Dialysis, or Persistent Decline in Kidney Function, Comparing Intravenous Sodium Bicarbonate With Intravenous Sodium Chloride.
Description: Death will be based on medical record and/or vital status registry documentation Need for acute dialysis will be defined as the initiation of any modality of renal replacement (intermittent hemodialysis, peritoneal dialysis, continuous renal replacement therapy, or sustained low-efficiency dialysis) Persistent decline in kidney function will be defined as an increase in serum creatinine of at least 50% from the baseline value collected pre-angiography to the measurement taken 90 days following the angiography.
Time Frame: Within 90 days following angiography
Measure: Count of Participants; unit: Participants
Groups:
- Sodium Bicarbonate: A grouping of participants receiving Sodium Bicarbonate.
- Saline: A grouping of participants receiving Saline.
Arm/Group | Sodium Bicarbonate | Saline
Number analyzed (Participants) | 2393 | 2379
Participants | 111 | 116
Statistical Analysis 1: Comparison: Sodium Bicarbonate vs Saline; Test type: Superiority; p = 0.70, Wald's Chi-Square; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.73 to 1.24]

2. Primary Outcome: Number of Participants With Serious, Adverse, Patient-Centered Events, Including Death, Need for Acute Dialysis, or Persistent Decline in Kidney Function, Comparing Oral N-Acetylcysteine With Oral Placebo.
Description: as for outcome 1
Time Frame: Within 90 days following angiography
Measure: Count of Participants; unit: Participants
Groups:
- N-Acetylcysteine (NAC): A grouping of participants receiving NAC.
- Placebo: A grouping of participants receiving placebo.
Arm/Group | N-Acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 2391 | 2381
Participants | 115 | 112
Statistical Analysis 1: Comparison: N-Acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.86, Wald's Chi-Square; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.78 to 1.34]

ADVERSE EVENTS:
Time Frame: Serious adverse events are collected from time of consent until 90 days post-angiography (per protocol). Adverse events were collected from time of consent until 35 days post-angiography (per protocol).
Description: All adverse events were collected regularly via developed case report forms and submitted electronically to the study electronic data capture (EDC) system. The definition for non-serious adverse events are derived from Veterans Health Administration (VHA) Handbook 1058.01, paragraph (a); The definition for serious adverse events are derived from VHA Handbook 1058.01, paragraph 4(r) and 21 Code of Federal Regulations (CFR) 312.32(a).
Groups:
- IV isotonic saline & oral placebo: IV isotonic saline and oral placebo drug capsule
  IV isotonic saline: The investigators will administer 3 ml/kg of isotonic saline over 1 hour at an infusion rate of not less than 1 mL/kg per hour and not more than 3 mL/kg per hour prior to the angiographic procedure, 1-1.5ml/kg per hour during angiography, and 6 ml/kg of isotonic saline over 4 hours following the procedure at an infusion rate of not less than 1 mL/kg per hour and not more than 1.5 mL/kg per hour. Providers will retain discretion to administer larger volumes of isotonic saline (up to a maximum of 12 mL/kg) over durations of up to 12 hours pre and 12 hours post-procedure.
  Placebo: A placebo study drug capsule will be administered orally 1 hour prior to angiography, 1 hour following the procedure, and then twice daily for the next 4 days.
- IV isotonic saline & oral N-acetylcysteine: IV isotonic saline and oral N-acetylcysteine drug capsule
  IV isotonic saline: The investigators will administer 3 ml/kg of isotonic saline over 1 hour at an infusion rate of not less than 1 mL/kg per hour and not more than 3 mL/kg per hour prior to the angiographic procedure, 1-1.5ml/kg per hour during angiography, and 6 ml/kg of isotonic saline over 4 hours following the procedure at an infusion rate of not less than 1 mL/kg per hour and not more than 1.5 mL/kg per hour. Providers will retain discretion to administer larger volumes of isotonic saline (up to a maximum of 12 mL/kg) over durations of up to 12 hours pre and 12 hours post-procedure.
  N-acetylcysteine: NAC will be administered at a dose of 1200mg orally 1 hour prior to angiography, 1 hour following the procedure, and then twice daily for the next 4 days.
- IV isotonic bicarbonate & oral placebo: IV isotonic bicarbonate and oral placebo drug capsule
  IV isotonic bicarbonate: The investigators will administer 3 ml/kg of isotonic bicarbonate over 1 hour at an infusion rate of not less than 1 mL/kg per hour and not more than 3 mL/kg per hour prior to the angiographic procedure, 1-1.5ml/kg per hour during angiography, and 6 ml/kg of isotonic bicarbonate over 4 hours following the procedure at an infusion rate of not less than 1 mL/kg per hour and not more than 1.5 mL/kg per hour. Providers will retain discretion to administer larger volumes of isotonic bicarbonate (up to a maximum of 12 mL/kg) over durations of up to 12 hours pre and 12 hours post-procedure.
  Placebo: A placebo study drug capsule will be administered orally 1 hour prior to angiography, 1 hour following the procedure, and then twice daily for the next 4 days.
- IV isotonic bicarbonate & oral N-acetylcysteine: IV isotonic bicarbonate and oral N-acetylcysteine drug capsule
  IV isotonic bicarbonate: The investigators will administer 3 ml/kg of isotonic bicarbonate over 1 hour at an infusion rate of not less than 1 mL/kg per hour and not more than 3 mL/kg per hour prior to the angiographic procedure, 1-1.5ml/kg per hour during angiography, and 6 ml/kg of isotonic bicarbonate over 4 hours following the procedure at an infusion rate of not less than 1 mL/kg per hour and not more than 1.5 mL/kg per hour. Providers will retain discretion to administer larger volumes of isotonic bicarbonate (up to a maximum of 12 mL/kg) over durations of up to 12 hours pre and 12 hours post-procedure.
  N-acetylcysteine: NAC will be administered at a dose of 1200mg orally 1 hour prior to angiography, 1 hour following the procedure, and then twice daily for the next 4 days.
Arm/Group | IV isotonic saline & oral placebo | IV isotonic saline & oral N-acetylcysteine | IV isotonic bicarbonate & oral placebo | IV isotonic bicarbonate & oral N-acetylcysteine
All-Cause Mortality (participants affected / at risk) | 28/1300 | 40/1292 | 33/1294 | 28/1291
Serious Adverse Events (participants affected / at risk) | 941/1300 | 1040/1292 | 1083/1294 | 941/1291
Other Adverse Events (participants affected / at risk) | 61/1300 | 158/1292 | 83/1294 | 170/1291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV isotonic saline & oral placebo (N=1300) | IV isotonic saline & oral N-acetylcysteine (N=1292) | IV isotonic bicarbonate & oral placebo (N=1294) | IV isotonic bicarbonate & oral N-acetylcysteine (N=1291)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 14 (15) | 10 (11) | 14 (15) | 15 (18)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 4 (5) | 2 (2)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 1 (2) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 8 (8) | 12 (12) | 2 (2) | 5 (6)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 19 (20) | 29 (32) | 27 (29) | 19 (20)
Angina pectoris (Cardiac disorders) | 7 (7) | 10 (10) | 6 (8) | 5 (6)
Angina unstable (Cardiac disorders) | 4 (4) | 14 (14) | 6 (6) | 12 (18)
Aortic valve disease (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Aortic valve disease mixed (Cardiac disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 2 (2) | 2 (2) | 4 (4) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 41 (44) | 47 (52) | 48 (52) | 47 (47)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 29 (33) | 32 (32) | 30 (31) | 26 (28)
Atrial flutter (Cardiac disorders) | 4 (4) | 5 (5) | 1 (1) | 6 (6)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 2 (2) | 3 (3) | 2 (2)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 3 (3) | 4 (4) | 1 (1)
Bradycardia (Cardiac disorders) | 5 (5) | 6 (6) | 4 (4) | 4 (5)
Bundle branch block left (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 4 (4) | 4 (4) | 3 (3) | 6 (6)
Cardiac failure acute (Cardiac disorders) | 4 (4) | 11 (11) | 8 (8) | 6 (7)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 37 (46) | 51 (57) | 61 (70) | 41 (48)
Cardiac perforation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 2 (2) | 2 (3) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 4 (4) | 3 (3) | 3 (3) | 6 (6)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 4 (4)
Cardiorenal syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiovascular deconditioning (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cor pulmonale (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 163 (186) | 178 (198) | 189 (213) | 145 (159)
Coronary artery dissection (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Coronary artery perforation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 8 (8) | 4 (4) | 7 (7) | 4 (4)
Coronary artery thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary ostial stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Degenerative mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 3 (3) | 4 (4) | 5 (5) | 4 (4)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Microvascular coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 7 (7) | 9 (9) | 11 (14) | 7 (7)
Mitral valve prolapse (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Myocardial infarction (Cardiac disorders) | 2 (2) | 6 (6) | 3 (3) | 11 (11)
Myocardial ischaemia (Cardiac disorders) | 6 (6) | 6 (6) | 3 (3) | 9 (11)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 4 (4) | 0 (0) | 2 (2)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rheumatic heart disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Sinus arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 5 (5) | 2 (2) | 2 (2) | 2 (2)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 6 (6) | 7 (8) | 9 (10) | 5 (5)
Bicuspid aortic valve (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Von Willebrand's disease (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acquired oesophageal web (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coeliac artery compression syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colonic pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral hernia incarcerated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 3 (4) | 5 (5) | 5 (5)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal mass (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (3)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal rupture (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic failure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (4) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Adverse drug reaction (General disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 4 (5) | 2 (2) | 3 (4) | 1 (1)
Catheter site haemorrhage (General disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 6 (6) | 10 (10) | 10 (10) | 7 (7)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Drug intolerance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 7 (7) | 2 (3) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulcer haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular stent restenosis (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Vascular stent thrombosis (General disorders) | 2 (4) | 1 (1) | 0 (0) | 1 (1)
Vessel puncture site thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (4)
Chronic hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cryptogenic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Gallbladder enlargement (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Hepatic congestion (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contrast media reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Selective IgA immunodeficiency (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Cardiac valve vegetation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 9 (9) | 7 (7) | 8 (8) | 8 (9)
Cellulitis gangrenous (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Clostridium bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Coccidioidomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Diabetic foot infection (Infections and infestations) | 2 (3) | 0 (0) | 2 (2) | 2 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterobacter pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Extradural abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 4 (4) | 3 (3) | 1 (1) | 1 (1)
Gas gangrene (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (3) | 2 (2) | 3 (3)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Graft infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Groin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemophilus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Incision site cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 2 (3)
Infected cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mediastinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 8 (8) | 8 (10) | 6 (7) | 2 (2)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 24 (25) | 21 (24) | 24 (27) | 18 (19)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 5 (6) | 5 (6) | 4 (5) | 4 (4)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 6 (6) | 6 (7) | 7 (9) | 5 (5)
Septic shock (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Serratia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serratia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 1 (2)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 8 (9) | 11 (13) | 14 (14) | 6 (8)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Viral diarrhoea (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 6 (7) | 1 (1)
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Arteriovenous graft aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Cerebral hyperperfusion syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 4 (4) | 6 (6) | 7 (8)
Fat embolism (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inappropriate schedule of drug administration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incision site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incorrect route of drug administration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peroneal nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Post procedural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 2 (3) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 5 (5) | 1 (1)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural stroke (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Postoperative fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Procedural hypertension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 0 (0) | 2 (2)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radiation proctitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transplant dysfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 3 (3) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anticoagulation drug level below therapeutic (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase MB increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram ST segment elevation (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left ventricular end-diastolic pressure increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary arterial wedge pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (3) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 0 (0) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 7 (8) | 3 (3)
Gout (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 4 (5) | 2 (2)
Hyperinsulinaemic hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2) | 3 (3) | 5 (5) | 6 (6)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 3 (6)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small cell lung cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 1 (3) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 12 (14) | 7 (7) | 4 (4) | 10 (11)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 7 (9) | 6 (6) | 8 (8) | 6 (6)
Cervical myelopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Movement disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nerve root compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Radicular pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 4 (4) | 7 (7)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 0 (0) | 2 (3) | 3 (3)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uraemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 4 (4) | 3 (3) | 1 (1) | 1 (1)
Delirium tremens (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Drug use disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Panic attack (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychiatric decompensation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Substance use disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 41 (43) | 67 (81) | 73 (88) | 58 (76)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder mass (Renal and urinary disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Bladder outlet obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 4 (4) | 3 (3) | 2 (3) | 3 (3)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 3 (3) | 4 (4) | 2 (2)
Nephropathy toxic (Renal and urinary disorders) | 3 (3) | 3 (3) | 3 (3) | 3 (4)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal artery occlusion (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Renal tubular necrosis (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary fistula (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 4 (4) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 1 (1) | 3 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 4 (4)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 14 (16) | 16 (19) | 9 (10)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 4 (4) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 10 (11) | 9 (11) | 8 (11)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 3 (4) | 4 (4)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2) | 6 (6) | 6 (7)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5) | 5 (5) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tonsillar ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 (7) | 1 (1) | 3 (5) | 2 (2)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcohol detoxification (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic valve replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arterial ligation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder catheterisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter management (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dialysis (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Drug therapy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot amputation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune tolerance induction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intra-aortic balloon placement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leg amputation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nutritional supplementation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parenteral nutrition (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Preoperative care (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prophylaxis (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal decompression (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombolysis (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toe amputation (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound drainage (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Air embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angiodysplasia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 4 (4) | 6 (6) | 5 (5) | 4 (4)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 6 (8) | 2 (2) | 2 (2) | 2 (2)
Dry gangrene (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Essential hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral artery dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 4 (4) | 2 (2) | 5 (5) | 2 (2)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 3 (3) | 5 (5) | 2 (2)
Hypertensive crisis (Vascular disorders) | 5 (5) | 1 (1) | 7 (7) | 4 (4)
Hypertensive emergency (Vascular disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Hypoperfusion (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 7 (7) | 7 (7) | 8 (9) | 11 (11)
Iliac artery occlusion (Vascular disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Labile hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurogenic shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 6 (6) | 2 (2) | 2 (2) | 8 (8)
Peripheral arterial occlusive disease (Vascular disorders) | 11 (12) | 9 (10) | 3 (3) | 12 (12)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Peripheral artery dissection (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Peripheral embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 5 (5)
Peripheral vascular disorder (Vascular disorders) | 8 (10) | 3 (3) | 7 (7) | 7 (7)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Shock (Vascular disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subclavian steal syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Temporal arteritis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV isotonic saline & oral placebo (N=1300) | IV isotonic saline & oral N-acetylcysteine (N=1292) | IV isotonic bicarbonate & oral placebo (N=1294) | IV isotonic bicarbonate & oral N-acetylcysteine (N=1291)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear Discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual Impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 7 (7) | 14 (14) | 12 (12)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 40 (40) | 4 (4) | 47 (48)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Frequent Bowel Movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Functional Gastrointestinal Disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 3 (3)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (9) | 31 (31) | 15 (15) | 28 (28)
Oesophageal Irritation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 11 (12) | 9 (9) | 10 (10)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site phlebitis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Infusion site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Sensation of foreign body (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural oedema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural hypertension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular end-diastolic pressure increased (Investigations) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 2 (2) | 2 (2)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 8 (8) | 0 (0) | 3 (3)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 2 (2) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 2 (2) | 6 (6)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"Cooperative Studies Program (CSP) retains ownership rights to all data collected in a CSP study…policies for data analysis and dissemination of results apply to all members of the Study Group (Study Chair (SC), Site Investigators (SIs), Study Biostatistician or Epidemiologist, etc.). If a SC or SI misuses study data, submits unauthorized manuscripts for publication, or releases results prior to the lifting of any embargoes or agreed upon time...administrative actions may be taken…"

DOCUMENTS (2):
  • Study Protocol (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT01467466/Prot_002.pdf
  • Statistical Analysis Plan (2016-08-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT01467466/SAP_001.pdf